CLINICAL TRIAL: NCT02687321
Title: The Role of HE4 in the Follow-up of Advanced Ovarian, Fallopian Tube and Primary Peritoneal Cancer: First Prospective Multicentre Observational Study
Brief Title: The Role of HE4 in the Follow-up of Advanced Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: University Hospital Pilsen (Other)
Responsible Party: Principal Investigator, Vit Weinberger, M.D., Ph.D., Brno University Hospital
Other Study IDs: HE4
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Advanced ovarian cancer patients: Patient with histologically confirmed advanced (FIGO III and IV) epithelial ovarian, fallopian tube or primary peritoneal carcinoma with complete remission after first line treatment are included into the study. The patient is regularly followed up every 3-4 months, blood sample collection is performed to determinate tumor marker found in blood, elevated by the presence of cancer recurrence. In case of one or both of tumor markers are elevated, computed tomography examination with intravenous contrast agent of chest and abdomen is performed to detect the recurrence of the disease.
  Interventions: Other: Determination of CA 125 and HE4, Computed tomography

INTERVENTIONS:
Other: Determination of CA 125 and HE4, Computed tomography — Blood sample collection to determinate tumor marker found in blood elevated by the presence of cancer recurrence.In case of one or both of tumor markers are elevated, computed tomography examination with intravenous contrast agent of chest and abdomen is performed to detect the recurrence of the disease.

SUMMARY:
To evaluate and to compare the effectiveness of CA-125 and HE4 serum levels in epithelial ovarian cancer (OC) in follow-up in terms of time to detection of elevation after the end of the first line treatment. To evaluate the lead-time of the rise of marker levels before epithelial OC recurrence diagnosis by Computed tomography (CT) imaging method. To evaluate the appropriate HE4 cut-off value for follow-up of patients after the treatment of ovarian, Fallopian tube and primary peritoneal cancer.

DETAILED DESCRIPTION:
Ovarian cancer (OC) is the second most common gynaecologic cancer and the leading cause of death from gynaecologic malignancy among women in industrialized countries. The global incidence in both developed and developing countries can be estimated as 165,000 new cases per year. A heavy difference in prognosis exists between the early-stage disease FIGO I-II (International Federation of Gynaecology and Obstetrics and the advanced stages (FIGO III-IV). Unfortunately, at present, we do not have an effective screening strategy for this malignancy; most (70-80%) of the cases are diagnosed as advanced-stage disease, and this explains the high mortality rate. These aggressive features of the OC encouraged in recent years a big effort in order to find new strategies for early diagnosis of OC. These studies focused dominant on new markers and diagnostic algorithms among new markers. HE4 is one of the most promising. It is a protein initially identified in the epithelium of the distal epididymis and may be involved in sperm maturation. Despite its wide distribution, it is overexpressed only in pathological tissue, and it has demonstrated good sensitivity and specificity in detecting OC, overcoming the traditional role of CA-125. Despite an aggressive upfront treatment strategy (surgery plus chemotherapy), leading to clinical remission in more than 80% of patients, the relapse-free survival varies from 95.8% (for early FIGO stages) to 33.6% (for advanced stages) at 2 years. At present, periodical evaluation of CA-125 combined with physical examination is the recommended strategy for OC follow-up, typically every 3 to 4 months in the first 2 years after primary treatment and then every 6 months until the fifth year. Five years' overall survival rate, however, is 49.7% (ranging from 83%-89% in stage I OC to 18% in stage IV). New markers should be tested in the follow-up of patients with OC to improve the surveillance program performance: the challenge is to try to anticipate the diagnosis of OC recurrence and to translate this early diagnosis of relapse in a survival improvement. Few studies only are available to date about HE4 use in follow up of ovarian cancer. All of these studies analyzed a small number of women (8-73). HE4 was shown as an earlier indicator of recurrence of OC with respect to CA-125, with a lead-time of 5 to 8 months. Only 1 prospective controlled study has been published. In this study the sensitivity and specificity of HE4, alone or in association with other markers (CA-125, CA-72-4), seems to be higher in the diagnosis of the OC relapse with respect to CA-125 alone. The other side of the question is whether the patient is advantaged by an earlier detection of the recurrent disease, in terms of overall survival, disease-free survival, and quality of life. Early detection and treatment of cancer in general or its recurrence are usually associated with better outcomes for patient, this being the rationale behind screening programs and follow-up strategies. In OC follow-up, periodical CA-125 evaluation can detect recurrence of cancer about 5 months before clinical signs or symptoms. At the same time, we have to remind, that treatments of relapsing OC are rarely curative and have heavy adverse effects, and elevation of CA-125 is often cause of anxiety in patients undergoing follow-up. The main study, that tried to clarify the role of CA-125 in OC follow-up was MRC OV05/EORTC (European Organisation for Research and Treatment of Cancer) 55955 trial a randomized study comparing early versus delayed treatment in women with relapsed OC. Patients in the delayed treatment group were treated only at clinical or symptomatic relapse. Women assigned to early treatment started chemotherapy 4.8 months earlier than those allocated to the delayed treatment. With a median follow-up of 56.9 months, there was no evidence of a difference in overall survival between the 2 groups. In particular, the results provided no evidence of an improved overall survival or a better quality of life in the early treatment group. The authors' explanation for these findings was that the lead-time between CA-125 rise and the clinical recurrence could be too short for chemotherapy to give a beneficial effect. At present, periodical evaluation of CA-125 combined with physical examination is the recommended strategy for OC follow-up, typically every 3 to 4 months in the first 2 years after primary treatment and then every 6 months until the fifth year. Five years' overall survival rate, however, is 49.7% (ranging from 83%-89% in stage I OC to 18% in stage IV).

ELIGIBILITY:
Inclusion Criteria:

* advanced ovarian cancer, stage FIGO III and IV
* histology types: high-grade serous, low-grade serous, endometrioid, clear cell, undifferentiated
* completed ovarian cancer surgery and platinum-based chemotherapy

Exclusion Criteria:

* positivity of tumor markers CA 125 and HE4 during study enrollment
* signs of cancer at computed tomography scan during study enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with histologically confirmed advanced epithelial ovarian, fallopian tube or primary peritoneal carcinoma with complete remission after first line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Serum levels of tumor marker CA-125 | two years after study enrollment
  kU/l
Serum levels of tumor marker HE4 | two years after study enrollment
  pmol/l

SECONDARY OUTCOMES:
Ovarian cancer recurrence diagnosed by computed tomography scan | two years after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Vit Weinberger, M.D., Ph.D., Principal Investigator — University Hospital Brno; Jiri Presl, M.D., Ph.D., Principal Investigator — University Hospital Pilsen
Locations (20):
- Czechia (7):
  - Brno University Hospital, Brno
  - Hospital Ceske Budejovice, České Budějovice
  - Faculty Hospital in Hradec Králové, Hradec Králové
  - Hospital Jihlava, Jihlava
  - Faculty Hospital Pilsen, Pilsen
  - General Hospital Prague, Prague
  - Regional Hospital Pilsen, Zlín
- University of Derecen, Debrecen, Hungary
- Poland (6):
  - Swietokrzyskie Cancer Center, Kielce
  - Cancer Center, M.Sklodowska-Curie Memorial Institute, Krakow
  - Medical University of Lublin, Lublin
  - Pomeranian Medical University, Szczecin
  - Medical University of Warsaw, Warsaw
  - Lower Silesian Cancer Center, Wroclaw
- Slovakia (4):
  - Institute of Oncology, Bratislava, Bratislava
  - National Institute of Oncology, Bratislava, Bratislava
  - University Hospital Bratislava, Bratislava
  - FN Trencín, Trenčín
- La Paz University Hospital. Madrid, Madrid, Spain
- Lviv State Regional Oncological Center, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No